CLINICAL TRIAL: NCT01977222
Title: Improving Functional Capacity in Fontan Patients Through Inspiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Fred Wu, Assistant in Cardiology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00006063
Record Dates: First submitted 2013-10-25; First posted 2013-11-06 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Congenital Heart Disease; Single Ventricle
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER (Experimental)
  Interventions: Device: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER

INTERVENTIONS:
Device: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER — Subjects will be provided with noseclips and a threshold impedance device set to 40% of their measured maximal inspiratory pressure and will be trained on using the device. Specifically, subjects will be instructed to breathe through the inspiratory muscle training device while wearing noseclips at a rate of 12 to 16 breaths per minute for 30 minutes a day, 5 days a week for 12 consecutive weeks. Each subject will be provided a customized schedule for increasing resistance by 2 cm H2O every 2 weeks to a maximum resistance of 41 cm H2O.

SUMMARY:
Mechanisms that typically result in increased cardiac output, such as inotropic support, increased heart rate, and decreased afterload, have a blunted effect in Fontan circulation. The "thoracic pump" is a contributor to venous return that has been largely unexplored in patients with Fontan physiology. Inspiratory muscle training can improve the performance of competitive athletes across a range of sports and can improve quality of life and functional capacity in heart failure patients, presumably by reducing inspiratory muscle fatigue and possibly by improving peripheral blood flow during exercise. One could surmise that the effects of these changes would be particularly important in the Fontan population. The investigators propose to study the effects of inspiratory muscle training on exercise and pulmonary function parameters in a cohort of adult Fontan patients.

The investigators hypothesize that a 12-week program of inspiratory muscle training with an inspiratory impedance threshold device will improve inspiratory muscle strength and endurance, and that this will translate into improved exercise performance in patients with Fontan physiology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Fontan physiology
* Undergoing cardiopulmonary stress testing
* Able to complete a previous cardiopulmonary stress test in the preceding 24 months
* Ability to comply with the inspiratory muscle training protocol
* Ability to return for repeat stress testing and pulmonary function testing 12 weeks after enrollment
* Ability to provide informed consent

Exclusion Criteria:

* Status post cardiac transplantation
* Current pregnancy or plans to become pregnant within the next 3 months (for females of childbearing potential)
* Active respiratory infection
* Active cigarette smoker
* Baseline oxygen saturation <90% at the previous clinic visit or exercise test
* Forced expired volume in 1 s and/or vital capacity <60% of predicted at the previous exercise test
* Cardiac surgery or catheter-based procedure in the preceding 18 months or planned surgery or catheter-based procedure within the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Wu, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive adult patients (≥18years old) with Fontan physiology were recruited through the outpatient cardiology clinic at Boston Children's Hospital between April 2014 and December 2014.
Pre-assignment Details: One subject who was enrolled and consented dropped out during the initial assessment due to inability to tolerate the metabolic cart during baseline exercise testing.
Period: Overall Study
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Only subjects who were subject to the intervention (inspiratory muscle training) are included
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Age at Fontan completion [Mean (Standard Deviation); unit: years] | 10.7 (8.0)
Fontan type [Count of Participants; unit: Participants]
  Lateral tunnel | 7
  Extracardiac conduit | 1
  Atriopulmonary connection | 3
Maximum inspiratory pressure [Mean (Standard Deviation); unit: cmH2O] | 87.7 (33.0)
Peak work rate [Mean (Standard Deviation); unit: Watts] | 116.5 (45.0)
Peak relative VO2 [Mean (Standard Deviation); unit: ml/kg/min] | 22.2 (8.0)
Peak relative VO2 [Mean (Standard Deviation); unit: % predicted] | 68.1 (14.3)
VE/VCO2 slope (ratio) [Mean (Standard Deviation); unit: ratio] | 34.1 (6.7)
Peak VE [Mean (Standard Deviation); unit: L/min] | 74.3 (27.8)
Peak heart rate [Mean (Standard Deviation); unit: beats per minute] | 132.3 (31.8)
Peak tidal volume [Mean (Standard Deviation); unit: L] | 2.03 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak VO2 Between Baseline and Post-inspiratory Muscle Training Measurements.
Time Frame: Baseline and after 12 weeks of training
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 11
ml/kg/min | 24.0 (9.8)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = 0.1673, t-test, 2 sided

2. Secondary Outcome: Change in Innocor Measurement (Inert Gas Rebreathing Method) of Cardiac Output at Peak Exercise
Time Frame: 12 weeks
Population: One individual failed to sustain maximal exercise long enough to complete measurement of cardiac output on her post-intervention study. That individual was therefore left out of the data analysis for cardiac output at peak exercise ONLY.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 10
L/min | 6.8 (1.9)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = 0.5745, t-test, 2 sided

3. Secondary Outcome: Change in SF-36 Health Survey Score (Physical Component Summary)
Description: The 36-Item Short Form (SF-36) Health Survey is a disease-generic survey of an individual's perceived health status and health-related quality of life. There are eight scaled scores, which are the weighted sums of the questions in their section. Each scale is transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. These eight scales are then used to calculate (using a proprietary formula) two summary scores: the physical component score (PCS), representing the four physical health scales (physical functioning, role physical, bodily pain, general health), and the mental component score (MCS), representing the four mental health scales (mental health, role emotional, vitality, social functioning). Component scores are norm-based with a mean of 50 (standardized to the US population) and a standard deviation of 10.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 11
units on a scale | 50.4 (9.8)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = .511, t-test, 2 sided

4. Other Pre Specified Outcome: Change in Maximum Voluntary Ventilation
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 10
L/min | 113.4 (31.5)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = 0.776, t-test, 2 sided

5. Other Pre Specified Outcome: Change in Maximal Inspiratory Pressure
Time Frame: Baseline and after 12 weeks of training
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 11
cmH2O | 96.0 (33.1)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = 0.5374, t-test, 2 sided

6. Other Pre Specified Outcome: Change in Oxygen Pulse at Peak Exercise
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 11
mL/beat | 13.1 (2.5)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = 0.3385, t-test, 2 sided

7. Other Pre Specified Outcome: Change in Peak Work Rate During Exercise
Time Frame: Baseline and after 12 weeks of training
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 11
Watts | 126.8 (47.0)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = 0.0189, t-test, 2 sided

8. Other Pre Specified Outcome: Change in VE/VCO2 Slope (Ratio) During Exercise
Time Frame: Baseline and after 12 weeks of training
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
Number analyzed (Participants) | 11
ratio | 31.4 (3.6)
Statistical Analysis 1: Comparison: THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER; Test type: Other; p = 0.1183, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Through completion of follow-up testing (completion of study), typically 12 weeks but no more than 15 weeks.
Description: Patients were contacted regularly throughout the training period by phone or email to evaluate for potential adverse events.
Arm/Group | THRESHOLD(TM) INSPIRATORY MUSCLE TRAINER
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
This pilot study was based on a limited number of patients. In addition, there was incomplete compliance with the prescribed inspiratory muscle training regimen. Finally, our subjects were relatively healthy and mostly had normal MIP at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes